CLINICAL TRIAL: NCT01058421
Title: Randomized Trial of Intensive Physical Therapy for Patients With Acute Respiratory Failure
Brief Title: Treatment of Critical Illness Polyneuromyopathy
Acronym: Do-It-Now
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0214
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Acute Respiratory Failure
Keywords: mechanical ventilation; acute respiratory failure; physical therapy; critical illness neuropathy; critical illness myopathy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive physical therapy (Experimental): four week intervention of daily intensive physical therapy
  Interventions: Procedure: intensive physical therapy
- control group (Active Comparator)
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: intensive physical therapy — four week course of daily intensive physical therapy
  Arms: Intensive physical therapy
Procedure: control group — four weeks of routine physical therapy
  Arms: control group

SUMMARY:
Acute respiratory failure is a heterogeneous disorder that results in more than 300,000 Americans requiring admission to an intensive care unit for invasive mechanical ventilatory support each year. Though acute respiratory failure is a pulmonary disorder, patients who survive their hospitalization are not limited by respiratory symptoms after discharge. Rather persistent neuromuscular weakness is the primary disorder that adversely alters their quality of life and ability to function on a daily basis. In this application the investigators plan to conduct a randomized clinical trial called the Do It Now study (Diagnosis and Treatment of Neuromuscular Weakness) to determine the effectiveness of an intensive physical therapy program for patients recovering from acute respiratory failure. This trial will establish the efficacy of the physical therapy programs that is currently performed for patients with acute respiratory failure in a non-evidence based manner across the United States.

DETAILED DESCRIPTION:
Acute respiratory failure is a heterogeneous disorder that results in more than 300,000 Americans requiring admission to an intensive care unit for invasive mechanical ventilatory support each year. Though acute respiratory failure is a pulmonary disorder, patients who survive are not limited by respiratory symptoms after discharge. Rather persistent neuromuscular weakness is the primary disorder that adversely affects their quality of life and ability to function on a daily basis. Weakness in these survivors is related to the development of critical illness polyneuromyopathy (CIPNM). Presently, there are no therapies to treat the estimated 110,000 acute respiratory failure survivors who have developed CIPNM each year. Based on the results of our national surveys of physical therapists and intensive care physicians, the utilization and types of physical therapy for patients recovering from acute respiratory failure with neuromuscular weakness varies significantly depending on the type of hospital and primary diagnosis of the patient. The investigators plan to perform a randomized clinical trial to determine the effectiveness of an intensive four week physical therapy program for patients with acute respiratory failure. This trial will determine the efficacy of the physical therapy programs that is currently performed in a non-evidence based manner for patients with acute respiratory failure across the United States. If successful, this study will pave the way for a larger multi-center clinical trial of intensive physical therapy for survivors of acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure requiring mechanical ventilation for at least four days.

Exclusion Criteria:

* Recent myocardial infarction within the last 3 weeks, presence of signs or symptoms of unstable angina or history of unstable arrhythmias including ventricular tachycardia and atrial fibrillation (HR > 100 bpm).
* Recent history of pulmonary embolism within the last six weeks.
* History of severe aortic stenosis.
* Presence of a dissecting aortic aneurysm.
* Significant language barrier that would limit the ability to participate in the physical therapy program.
* Patients who live greater than 45 miles from the University of Colorado Hospital.
* Underlying disorder that makes it unlikely that the patient will survive 6 months.
* Severe physical or cognitive impairment that would impair their ability to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, M.D., Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Anthony Hospital, Lakewood, Colorado

IPD SHARING:
Plan to Share IPD: Yes
We have created a de-identified data set that is available to other investigators upon request.

REFERENCES:
- [Derived] Neumeier A, Nordon-Craft A, Malone D, Schenkman M, Clark B, Moss M. Prolonged acute care and post-acute care admission and recovery of physical function in survivors of acute respiratory failure: a secondary analysis of a randomized controlled trial. Crit Care. 2017 Jul 21;21(1):190. doi: 10.1186/s13054-017-1791-1. PMID 28732512
- [Derived] Moss M, Nordon-Craft A, Malone D, Van Pelt D, Frankel SK, Warner ML, Kriekels W, McNulty M, Fairclough DL, Schenkman M. A Randomized Trial of an Intensive Physical Therapy Program for Patients with Acute Respiratory Failure. Am J Respir Crit Care Med. 2016 May 15;193(10):1101-10. doi: 10.1164/rccm.201505-1039OC. PMID 26651376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Deceased subjects were removed from starting period subject numbers for subsequent outcome periods in each cohort. All non-deceased subjects were included in period outcomes analysis and categorized as death in subsequent period, lost to follow-up, remained in hospital or other facility.
Groups:
- Intensive Physical Therapy Treatment Group: Participants received intensive physical therapy 7 days per week, and outpatient physical therapy 3 days per week, beginning Day 1 through Day 28.
- Standard of Care Physical Therapy Group: Participants received standard of care inpatient physical therapy 3 days per week, and no outpatient physical therapy, beginning Day 1 through Day 28.
Period: 1 Month Outcomes
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Started | 59 | 61
Completed | 20 | 19
Not Completed | 39 | 42
Not completed — Death | 10 | 6
Not completed — Lost to Follow-up | 8 | 7
Not completed — Remained in Hospital | 5 | 12
Not completed — Remained in Other Facility | 16 | 17
Period: 3 Month Outcomes
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Started (Deceased subjects were not included in subsequent Period beginning subject started totals.) | 49 (59 (Subjects started Period 1) minus 10 (deceased subjects during Period 1) = 49 started Period 2.) | 55 (61 (Subjects started Period 1) minus 6 (deceased subjects during Period 1) = 55 started Period 2.)
Completed | 29 | 29
Not Completed | 20 | 26
Not completed — Death | 3 | 5
Not completed — Lost to Follow-up | 12 | 11
Not completed — Remained in Hospital | 0 | 2
Not completed — Remained in Other Facility | 5 | 8
Period: 6 Month Outcomes
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Started (Deceased subjects were not included in subsequent Period beginning subject started totals.) | 46 (55 (subjects started Period 1) minus 13 (deceased subjects in Periods 1 & 2) = 46 started Period 3.) | 50 (61 (subjects started Period 1) minus 11 (deceased subjects in Periods 1 & 2) = 50 started Period 3.)
Completed | 27 | 24
Not Completed | 19 | 26
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 16 | 21
Not completed — Remained in Other Facility | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Median (Full Range); unit: years] | 56 [42 to 70] | 49 [34 to 64] | 53 [34 to 70]
Sex/Gender, Customized [Number; unit: participants]
  Female | 24 | 26 | 50
  Male | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Variable for This Study Will be the Short Form of the Continuous Scale Physical Functional Performance Test (CS-PFP) Called the PFP-10
Description: The CS-PFP-10 provides an overall score and scores for upper body strength, upper body flexibility, lower body strength, balance and coordination, and endurance. The test is used to assess an individual's overall capacity to carry out activities of daily living by measuring and quantifying 10 typical activities including sweeping a floor, transferring clothes from a washer to a dryer, and carrying groceries. Tasks are quantified using time alone, time and weight, and distance. This test provides a realistic and practical measure of movement capacity and ability to accomplish sustained activity. CS-PFP-10 scores are scored from 0 to 100, with higher scores indicating better function. If patients remained in the hospital or in a long-term care facility a the time of assessment, then received a score of 0. All tests were conducted in a standardized physical therapy laboratory by a physical therapist formally trained in conducting the CS-PFP-10 and blinded to group/arm assignment.
Time Frame: 1 month
Population: 41 of 59 subjects were analyzed in the Intensive Treatment Group (20 completed outcomes testing + 5 remained in hospital + 16 remained in another facility = 41 subjects). 48 of 61 Standard of Care Group subjects were analyzed (19 completed outcomes testing + 12 remained in hospital + 17 remained in another facility = 48).
Measure: Mean (Standard Error); unit: score
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 41 | 48
score | 19.0 (3.7) | 20.9 (4.1)

2. Secondary Outcome: ICU-free Days
Description: Number of ICU-free days at Day 28.
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
Days | 13 [3 to 18] | 11 [4 to 18]

3. Secondary Outcome: ICU Length of Stay
Description: Median ICU length of stay through Day 28
Time Frame: Total Days through Day 28
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
Days | 15 [10 to 25] | 16 [10 to 24]

4. Secondary Outcome: Mechanical Ventilation Duration
Description: The total number of ventilated days from hospital admission to extubation, death or discharge over the complete duration of study participation, up to 180 days.
Time Frame: up to 180 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
Days | 10 [7 to 18] | 10 [7 to 19]

5. Secondary Outcome: Hospital Free Days
Time Frame: Through Day 28
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
Days | 7 [0 to 12] | 7 [0 to 14]

6. Secondary Outcome: Hospital Length of Stay
Description: The total number of hospital days during study participation, up to 180 days.
Time Frame: up to 180 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
Days | 21 [16 to 32] | 21 [14 to 38]

7. Secondary Outcome: Discharged to Home
Description: Percentage of subjects discharged to home from study hospital
Time Frame: Through Day 28
Measure: Number; unit: percentage of participants
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 59 | 61
percentage of participants | 51 | 49

8. Secondary Outcome: Institution Free Days
Description: Median number of days subjects were alive and free of hospitalization or living in a longer-term care, rehabilitation, or skilled nursing facility.
Time Frame: At Day 90
Population: Deceased subjects were not included in subsequent Period beginning subject started totals.
  59 (Subjects started Period 1) minus 10 (deceased subjects during Period 1) = 49 started Period 2.
  61 (Subjects started Period 1) minus 6 (deceased subjects during Period 1) = 55 started Period 2.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 49 | 55
Days | 61 [39 to 73] | 56 [33 to 75]

9. Secondary Outcome: Institution Free Days
Description: Median number of days subjects were alive and free of hospitalization or living in a long-term care, rehabilitation, or skilled nursing facility.
Time Frame: Day 180
Population: Deceased subjects were not included in subsequent Period beginning subject started totals.
  55 (subjects started Period 1) minus 13 (deceased subjects in Periods 1 & 2) = 46 started Period 3.
  61 (subjects started Period 1) minus 11 (deceased subjects in Periods 1 & 2) = 50 started Period 3.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Number analyzed (Participants) | 46 | 50
Days | 151 [129 to 163] | 146 [123 to 165]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intensive Physical Therapy Treatment Group | Standard of Care Physical Therapy Group
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 1/59 | 1/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Physical Therapy Treatment Group (N=59) | Standard of Care Physical Therapy Group (N=61)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — One subject had a syncopal episode during a physical therapy session.
Polyarthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One subject was readmitted to study hospital for 2 day stay after initial hospital stay due to polyarthralgia that was possibly related to physical therapy interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No